CLINICAL TRIAL: NCT04816201
Title: Electroacupuncture to Assist Ventilator Weaning in Severe Stroke: a Randomized, Sham-controlled Pilot Study
Brief Title: Electroacupuncture to Assist Ventilator Weaning in Severe Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fang Yuan, PhD, MD, The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZF2021-035
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Severe Stroke; Electroacupuncture
Keywords: ventilator weaning; severe stroke; electroacupuncture
MeSH Terms: conditions — Stroke | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): Participants in the electroacupuncture group received acupuncture at Xuanji (CV21), Danzhong (CV27), Qihai (CV06), Guanyuan (CV04), and bilateral Liangmen (ST21) and Zusanli (ST36). After skin disinfection, sterile adhesive pads were placed on these acupoints, and acupuncture needles were inserted through the adhesive pads approximately 50 to 60 mm into the skin. Paired electrodes from the electroacupuncture apparatus were attached to the needle handles of Xuanji (CV21) and Danzhong (CV27), Qihai (CV06), Guanyuan (CV04), bilateral Liangmen (ST21), and bilateral Zusanli (ST36). The electroacupuncture stimulation lasted for 30 minutes with an intermittent wave of 50 Hz and a current intensity of 1 to 5mA (preferably with the skin around the acupoints shivering mildly without pain). Participants received 1 treatment session per day until the success of ventilator weaning (up to 21 days).
  Interventions: Other: Electroacupuncture
- Sham electroacupuncture (Sham Comparator): Participants in the sham electroacupuncture group received sham electroacupuncture with a pragmatic placebo needle on sham acupoints. The sham Xuanji (CV21) point was 1 cun (≈20 mm) above to Xuanji (CV21), the sham Danzhong (CV27) point was 1 cun(≈20mm) above to Danzhong (CV27), the sham Qihai (CV06) point was 1 cun(≈20mm) above to Qihai (CV06), the sham Guanyuan (CV04) point was 1 cun(≈20mm) above to Guanyuan (CV04), the sham Liangmen (ST21) point was 1 cun(≈20mm) lateral to Liangmen (ST21), and the sham Zusanli (ST36) point was 1 cun(≈20mm) lateral to Zusanli (ST36). Procedures, electrode placements, and other treatment settings were the same as in the electroacupuncture group but with no skin penetration or electricity output.
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Electroacupuncture at Xuanji (CV21), Danzhong (CV27), Qihai (CV06), Guanyuan (CV04), and bilateral Liangmen (ST21) and Zusanli (ST36).

SUMMARY:
The purpose of this study is to evaluate the efficacy of electroacupuncture in assisting ventilator weaning in patients with severe stroke

DETAILED DESCRIPTION:
Disuse atrophy of the major respiratory muscles and diaphragmatic dysfunction often develop during mechanical ventilation, and cause difficulties in ventilator weaning. Electroacupuncture was indicated to promote activities of diaphragm and improve diaphragmatic function. Our aim is to evaluate the efficacy of electroacupuncture in assisting ventilator weaning in patients with severe stroke. 100 eligible patients will be randomly assigned to receive electroacupuncture or sham electroacupuncture treatment one session per day until the success of ventilator weaning (up to 21 days). The primay outcome is the ventilation duration within 21 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years and ≤ 75 years ;
2. within 7 days after the onset of stroke (ischemic or hemorrhagic), confirmed by a computed tomography (CT) or magnetic resonance imaging (MRI) scan of the brain;
3. GCS on admission ≤ 12 or NIHSS on admission ≥ 11 or APACHEⅡ ≥ 15;
4. received mechanical ventilation;
5. written informed consent is able to be obtained directly from the patient or an appropriate surrogate, based on local ethics committee recommendations.

Exclusion Criteria:

1. expected to be ventilated for < 24 h;
2. already ventilated for > 72 h;
3. GCS <5;
4. with unstable vital signs and requiring the use of vasoactive agents;
5. concomitant medical illness that would interfere with the outcome assessments and/or follow-up;
6. had spinal cord injury above T8 level, or lower motor neuron impairment, or neuromuscular junction impairment，or chest wall deformities, or chest wall injuries within 6 months, or chest or abdominal surgery within 4 week, or were pregnant;
7. had acute skin injury on the selected acupoints;
8. currently participating in other investigational trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ventilation duration | within 21 days after enrollment
  hours

SECONDARY OUTCOMES:
rate of successful ventilator weaning | within 21 days after enrollment
  percentage
diaphragm muscle thickness | on day 7, day 14 and day 21
  mm
diaphragm thickening fraction | on day 7, day 14 and day 21
  percentage
diaphragm excursion | on day 7, day 14 and day 21
  mm
rate of death | within 21 days after enrollment
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Wang, PhD, Study Director — The Second Affiliated Hospital of Guangzhou University of Chinese Medicine
Locations (1):
- The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The detailed datasets used and/or analyzed during the current study are available upon reasonable request.

REFERENCES:
- [Background] Tobin MJ, Laghi F, Jubran A. Ventilatory failure, ventilator support, and ventilator weaning. Compr Physiol. 2012 Oct;2(4):2871-921. doi: 10.1002/cphy.c110030. PMID 23720268
- [Background] Kim WY, Lim CM. Ventilator-Induced Diaphragmatic Dysfunction: Diagnosis and Role of Pharmacological Agents. Respir Care. 2017 Nov;62(11):1485-1491. doi: 10.4187/respcare.05622. Epub 2017 Jul 11. PMID 28698263
- [Background] Chen YJ, Hwang SL, Li CR, Yang CC, Huang KL, Lin CY, Lee CY. Vagal withdrawal and psychological distress during ventilator weaning and the related outcomes. J Psychosom Res. 2017 Oct;101:10-16. doi: 10.1016/j.jpsychores.2017.07.012. Epub 2017 Jul 29. PMID 28867413
- [Background] Ataya A, Silverman EP, Bagchi A, Sarwal A, Criner GJ, McDonagh DL. Temporary Transvenous Diaphragmatic Neurostimulation in Prolonged Mechanically Ventilated Patients: A Feasibility Trial (RESCUE 1). Crit Care Explor. 2020 Apr 29;2(4):e0106. doi: 10.1097/CCE.0000000000000106. eCollection 2020 Apr. PMID 32426748
- [Background] Essouri S, Baudin F, Mortamet G, Beck J, Jouvet P, Emeriaud G. Relationship Between Diaphragmatic Electrical Activity and Esophageal Pressure Monitoring in Children. Pediatr Crit Care Med. 2019 Jul;20(7):e319-e325. doi: 10.1097/PCC.0000000000001981. PMID 31107378
- [Background] Abdelwahed WM, Abd Elghafar MS, Amr YM, Alsherif SEI, Eltomey MA. Prospective study: Diaphragmatic thickness as a predictor index for weaning from mechanical ventilation. J Crit Care. 2019 Aug;52:10-15. doi: 10.1016/j.jcrc.2019.03.006. Epub 2019 Mar 15. No abstract available. PMID 30904733
- [Background] Bellani G, Bronco A, Arrigoni Marocco S, Pozzi M, Sala V, Eronia N, Villa G, Foti G, Tagliabue G, Eger M, Pesenti A. Measurement of Diaphragmatic Electrical Activity by Surface Electromyography in Intubated Subjects and Its Relationship With Inspiratory Effort. Respir Care. 2018 Nov;63(11):1341-1349. doi: 10.4187/respcare.06176. PMID 30389829
- [Background] McCaughey EJ, Jonkman AH, Boswell-Ruys CL, McBain RA, Bye EA, Hudson AL, Collins DW, Heunks LMA, McLachlan AJ, Gandevia SC, Butler JE. Abdominal functional electrical stimulation to assist ventilator weaning in critical illness: a double-blinded, randomised, sham-controlled pilot study. Crit Care. 2019 Jul 24;23(1):261. doi: 10.1186/s13054-019-2544-0. PMID 31340846
- [Background] McCaughey EJ, Berry HR, McLean AN, Allan DB, Gollee H. Abdominal Functional Electrical Stimulation to Assist Ventilator Weaning in Acute Tetraplegia: A Cohort Study. PLoS One. 2015 Jun 5;10(6):e0128589. doi: 10.1371/journal.pone.0128589. eCollection 2015. PMID 26047468